CLINICAL TRIAL: NCT03734497
Title: Carotid Flow Time Measurement Guided Fluid Management During Spinal Anesthesia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Ethical approval not obtained
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, DILEK YAZICIOGLU, Assoc Prof, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Spinal anesthesia-FTc
Record Dates: First submitted 2018-11-01; First posted 2018-11-08 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2021-09

CONDITIONS: Meniscus Disorder
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Prospective randomised
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group Control (Active Comparator): will receive 2 ml/kg "Ringer's lactate" Lafleks® during anesthesia
  Interventions: Other: Group Control 2 ml/kg "Ringer's lactate" Lafleks®
- Group Preloading (Experimental): will receive 10 ml/kg "Ringer's lactate" Lafleks® fluid preloading
  Interventions: Other: Group Preloading 10 ml/kg "Ringer's lactate" Lafleks®
- Group Carotis FTc (Experimental): will receive 500 ml "Ringer's lactate" Lafleks® if the patient is fluid responder
  Interventions: Other: Group Carotis FTc 500 ml "Ringer's lactate" Lafleks®

INTERVENTIONS:
Other: Group Carotis FTc 500 ml "Ringer's lactate" Lafleks® — will receive 500 ml "Ringer's lactate" Lafleks® if the patient is fluid responder
  Arms: Group Carotis FTc
Other: Group Preloading 10 ml/kg "Ringer's lactate" Lafleks® — will receive 10 ml/kg "Ringer's lactate" Lafleks® fluid preloading
  Arms: Group Preloading
Other: Group Control 2 ml/kg "Ringer's lactate" Lafleks® — will receive 2 ml/kg "Ringer's lactate" Lafleks® during anesthesia
  Arms: Group Control

SUMMARY:
Fluid management is a fundamental aspect of anesthesia. Several monitorization methods have been introduced to optimize fuid management.

To date neither of them were ideal. Corrected flow time measurement (FTc) in the carotid artery was recently introduced to detect fluid responsiveness.

Spinal anesthesia causes hypotension and fluid preloading is suggested to overcome this problem.

The aim of this study is to evaluate the effect of FTc guided fluid loading on spinal anesthesia induced hypotension.

DETAILED DESCRIPTION:
Patients will be randomly allocated into 3 groups. Group C (Control) will receive spinal anesthesia after initiation of intravenous (iv) access without fluid preloading and will receive 2 ml/kg Ringer's lactate during anesthesia..

Group P (preloading) will receive 10 ml/kg Ringer's lactate before spinal block.

In Group FTc, ultrasonographic measurement of corrected flow time in carotid artery will be measured using 10-5 megahertz linear probe. On the two-dimensional image, the optimal image of the long-axis view will be obtained at the left common carotid artery. The sample volume will be placed on the center of the lumen, 2 cm proximal to the bulb, and a pulsed wave Doppler examination will be performed. Cardiac cycle time and carotid flow time will be measured. Carotid flow time will be measured between the upstroke of the flow tracing and the dicrotic notch, and it will be corrected for pulse rate by dividing flow time by the square root of the cardiac cycle time to calculate corrected carotid artery flow time (flow time/√cycle time).

The blood pressure will be measured 5 minutes before spinal anesthesia is commenced (baseline) and every minute afterwards until end of surgery.

Group FTc will receive a 500 mL Ringer's lactate bolus if the FTc is <349 ms (fluid responder); the FTc measurement will be repeated 15 minutes later and additional 500 mL Ringer's lactate bolus will be applied if the patient is still considered fluid responder; this sequence will be repeated until the patient's FTc is > 349 ms (non responder).

Ephedrine bolus will be used in allh groups if the mean arterial pressure drops below 30% of the baseline value.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (19-80 years of age) who were scheduled to undergo arthroscopic knee surgery under spinal anesthesia

Exclusion Criteria:

* Mean blood pressure < 70 mmHg before induction of general anesthesia
* Patients who have currently taken angiotensin-converting enzyme inhibitor
* Patients who have currently taken angiotensin receptor blocker
* the presence of carotid artery stenosis > 50%
* cardiac rhythm other than sinus
* unstable angina
* a left ventricular ejection fraction of < 40%
* severe vascular disease
* implanted pacemaker/cardioverter
* autonomic nervous system disorders
* pregnancy

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07 (Estimated); Primary Completion 2022-09 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with Hypotension | 5 minutes after induction of spinal anesthesia
  Mean arterial pressure >30% lower than baseline value

SECONDARY OUTCOMES:
Number of patients receiving Vasopressor therapy | 5 minutes after induction of spinal anesthesia
  Ephedrine will be administered if mean arterial pressure drops >30% than baseline value

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Ünal, Principal Investigator — University of Health Sciences Dıskapı Yıldırım Beyazıt Training and Research Hospital
Locations (1):
- Diskapi Yildirim Beyazit Teaching and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee JE, George RB, Habib AS. Spinal-induced hypotension: Incidence, mechanisms, prophylaxis, and management: Summarizing 20 years of research. Best Pract Res Clin Anaesthesiol. 2017 Mar;31(1):57-68. doi: 10.1016/j.bpa.2017.01.001. Epub 2017 Jan 8. PMID 28625306
- [Result] Song Y, Kwak YL, Song JW, Kim YJ, Shim JK. Respirophasic carotid artery peak velocity variation as a predictor of fluid responsiveness in mechanically ventilated patients with coronary artery disease. Br J Anaesth. 2014 Jul;113(1):61-6. doi: 10.1093/bja/aeu057. Epub 2014 Apr 9. PMID 24722322
- [Result] Ceruti S, Anselmi L, Minotti B, Franceschini D, Aguirre J, Borgeat A, Saporito A. Prevention of arterial hypotension after spinal anaesthesia using vena cava ultrasound to guide fluid management. Br J Anaesth. 2018 Jan;120(1):101-108. doi: 10.1016/j.bja.2017.08.001. Epub 2017 Nov 23. PMID 29397116